CLINICAL TRIAL: NCT04603391
Title: An Assessment of the Drug Interaction Potential Between Oral Cannabidiol (Epidiolex®) and the CES1 Substrate Methylphenidate in Healthy Volunteers
Brief Title: Cannabidiol and CES1 Interactions in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Consortium for Medical Marijuana Clinical Outcomes Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB202002547-A; OCR39758 (Other: UF OnCore)
Record Dates: First submitted 2020-10-22; First posted 2020-10-26 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-06

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Cannabidiol; Methylphenidate

STUDY DESIGN:
Intervention Model Description: An open-label, randomized crossover design is proposed wherein healthy volunteer subjects (n=12) would receive a single dose of immediate-release dl-methylphenidate (Ritalin®) concomitantly with orally administered CBD (Epidiolex®) solution or an equal volume of Epidiolex® placebo solution (i.e vehicle with no CBD) which have been dosed to plasma steady-state conditions.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CBD, then placebo (Experimental): Subjects received a three day run in of CBD 750 mg orally twice daily (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]). On day four, all subjects returned to the clinical research center to receive one oral dose of CBD 750 mg (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
  After a minimum washout period of five days, subjects received a three day run in of 7.5 ml of Epidiolex® placebo solution (no CBD) orally twice daily. On day four, all subjects returned to the clinical research center to receive one oral dose of 7.5 mL of Epidiolex® placebo solution (no CBD) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
  Interventions: Drug: dl-Methylphenidate plus Cannabidiol; Drug: dl-Methylphenidate plus Cannabidiol Placebo solution
- Placebo, then CBD (Experimental): Subjects received a three day run in of 7.5 ml of Epidiolex® placebo solution (no CBD) orally twice daily. On day four, all subjects returned to the clinical research center to receive one oral dose of 7.5 mL of Epidiolex® placebo solution (no CBD) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
  After a minimum washout period of five days, subjects received a three day run in of CBD 750 mg orally twice daily (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]). On day four, all subjects returned to the clinical research center to receive one oral dose of CBD 750 mg (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
  Interventions: Drug: dl-Methylphenidate plus Cannabidiol; Drug: dl-Methylphenidate plus Cannabidiol Placebo solution

INTERVENTIONS:
Drug: dl-Methylphenidate plus Cannabidiol — Subjects will be administered one 10 mg tablet of dl-methylphenidate (Ritalin®) plus 7.5 mL Epidiolex® solution
  Other Names: Ritalin®; Epidiolex®
Drug: dl-Methylphenidate plus Cannabidiol Placebo solution — Subjects will be administered one 10 mg tablet of dl-methylphenidate (Ritalin®) plus 7.5 mL of Epidiolex® placebo solution
  Other Names: Ritalin®; Epidiolex®

SUMMARY:
The proposed study will assess the drug interaction potential between oral cannabidiol (Epidiolex®) and the carboxylesterase 1 (CES1) substrate methylphenidate (Ritalin®) in 12 healthy research subjects

DETAILED DESCRIPTION:
Cannabidiol (CBD) is a widely utilized nonpsychoactive cannabinoid available as an OTC supplement, a component of medical cannabis, and a prescriptive treatment of childhood epilepsies. In vitro studies suggest CBD may inhibit a number of drug-metabolizing enzymes, including carboxylesterase 1 (CES1). The aim of this study was to evaluate effect of CBD on the disposition of the CES1 substrate methylphenidate (MPH). This was a randomized, placebo-controlled, crossover study involving 12 healthy subjects. Each subject ingested 750 mg of CBD solution, or alternatively, a placebo solution twice daily for a 3-day run-in period followed by an additional CBD dose (or placebo) and a single 10 mg dose of MPH and completed serial blood sampling for pharmacokinetic analysis. MPH and CBD concentrations were measured by liquid chromatography with tandem mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Age: 21-45 years
* Gender: males and females (50:50)
* Race or ethnicity: no restrictions
* Body Mass Index (BMI) between 18.5 to 28 kg/m2 (inclusive)
* Satisfactory completion of the screening medical history, physical exam, and laboratory evaluations.
* Females of child-bearing potential must have a negative urine pregnancy test prior to enrollment and avoid pregnancy during study participation.
* With the exception of oral contraceptives, subjects must not be taking prescription or OTC medication for the duration of study participation
* Subjects must have no ongoing use of any botanical/nutritional supplement, vitamin, or energy drink for the duration of study participation

Exclusion Criteria:

* The presence of a known allergy, hypersensitivity, or adverse reaction to CBD or cannabis, or sesame seed oil
* The presence of a known allergy, hypersensitivity, or adverse reaction to methylphenidate or dexmethylphenidate (Focalin®)
* A history (within the past year) or presence of clinically significant cardiovascular, cerebrovascular, renal, hepatic, gastrointestinal, pulmonary, immunological, hematological, endocrine, or neurologic disease will render subjects ineligible for the study.
* The presence of any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion including;

  1. Gastric bezoar
  2. Swallowing disorders
  3. Strictures
  4. Fistulas
  5. GI obstruction
  6. Severe dsyphasgia
  7. Crohn's disease
  8. Diverticulitis
  9. A positive urine pregnancy test.
  10. A positive Urine Drug Screen
  11. Any concomitant prescription medication, OTC medication, herbal or other dietary supplement or vitamins during the study period.

All subjects must be medication-free from 7 Days before initiation of the first active study day, through the duration of the study. This exclusion the use of vitamins, herbal preparations and OTC supplements.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Markowitz, Pharm.D, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, subjects were assigned a screening visit date at the Clinical Research Center to obtain a medical history, physical, and routine lab tests including a complete blood count, comprehensive metabolic panel, urinalysis, and urine drug screen.
Groups:
- First Methylphenidate and CBD, Then Methylphenidate and Placebo: Subjects received a three day run in of CBD 750 mg orally twice daily (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]). On day four, all subjects returned to the clinical research center to receive one oral dose of CBD 750 mg orally (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
  After a minimum washout period of five days, subjects received a three day run in of 7.5 ml of Epidiolex® placebo solution (no CBD) orally twice daily. On day four, all subjects returned to the clinical research center to receive one oral dose of 7.5 mL of Epidiolex® placebo solution (no CBD) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
- First Methylphenidate and Placebo, Then Methylphenidate and CBD: Subjects received a three day run in of 7.5 ml of Epidiolex® placebo solution (no CBD) orally twice daily. On day four, all subjects returned to the clinical research center to receive one oral dose of 7.5 mL of Epidiolex® placebo solution (no CBD) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
  After a minimum washout period of five days, subjects received a three day run in of CBD 750 mg orally twice daily (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]). On day four, all subjects returned to the clinical research center to receive one oral dose of CBD 750 mg orally (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
Period: First Intervention (4 Days)
Arm/Group | First Methylphenidate and CBD, Then Methylphenidate and Placebo | First Methylphenidate and Placebo, Then Methylphenidate and CBD
Started | 8 | 6
Completed | 6 | 6
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Washout (Minimum 5 Days)
Arm/Group | First Methylphenidate and CBD, Then Methylphenidate and Placebo | First Methylphenidate and Placebo, Then Methylphenidate and CBD
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Second Intervention (4 Days)
Arm/Group | First Methylphenidate and CBD, Then Methylphenidate and Placebo | First Methylphenidate and Placebo, Then Methylphenidate and CBD
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Subjects for Both Sequences: Sequence 1: Subjects received a three day run in of 7.5 mL of Epidiolex® solution [100 mg/ml]). On day four, all subjects returned to the clinical research center to receive one oral dose of 7.5 mL of Epidiolex® solution [100 mg/ml]) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast). After a minimum washout period of five days, subjects received a three day run in of 7.5 ml of Epidiolex® placebo solution orally twice daily. On day four, all subjects returned to the clinical research center to receive one oral dose of 7.5 mL of Epidiolex® placebo solution and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
  Sequence 2: Subjects received a three day run in of 7.5 ml of Epidiolex® placebo solution orally twice daily. On day four, all subjects returned to the clinical research center to receive one oral dose of 7.5 mL of Epidiolex® placebo solution and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast). After a minimum washout period of five days, Subjects received a three day run in of 7.5 mL of Epidiolex® solution [100 mg/ml]). On day four, all subjects returned to the clinical research center to receive one oral dose of Epidiolex® solution [100 mg/ml]) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
Arm/Group | All Study Subjects for Both Sequences
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.67 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Differences in the Geometric Mean Ratio (GMR) of the Peak Concentration (Cmax) Will be Compared Between the Two Exposure Conditions; i.e. Methylphenidate + CBD vs Methylphenidate + Placebo.
Description: Plasma methylphenidate (MPH) concentrations for both arms were determined by using a liquid-liquid extraction method and LC-MS/MS analysis. Peak concentration (Cmax) was reported as observed for each subject. The geometric mean ratios (GMR) of the Cmax for MPH were compared between the two exposure conditions, i.e., MPH with CBD versus MPH with placebo. In brief, if the 90% confidence interval (CI) of GMR for Cmax between the CBD group and placebo group extend beyond the FDA's established bioequivalent limits of 0.8-1.25, the result was interpreted to represent a DDI. In our case, a GMR greater than 1.25 would be indicative of a DDI, since CBD would impair CES1's ability to efficiently metabolize MPH, thus a higher ratio of Cmax's of MPH in our CBD group relative to our placebo group.
Time Frame: 8 hours
Population: Each subject served as their own control, so since all 12 subjects that completed the study went through both arms, we were able to analyze the both arms for each subject. Hence, 12 subjects gave us 24 arms (2 arms/subject). The Cmax for each subject in the methylphenidate and CBD arm was directly compared to their methylphenidate and placebo arm, allowing us to determine the ratio of change in the presence of CBD.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Groups:
- All Participants: Methylphenidate and CBD Arm Only
  Subjects received a three day run in of CBD 750 mg orally twice daily (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]). On day four, all subjects returned to the clinical research center to receive one oral dose of CBD 750 mg orally (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
  Methylphenidate and Placebo Arm Only
  Subjects received a three day run in of 7.5 ml of Epidiolex® placebo solution (no CBD) orally twice daily. On day four, all subjects returned to the clinical research center to receive one oral dose of 7.5 mL of Epidiolex® placebo solution (no CBD) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
  The subsequent analysis compared the geometric mean ratio of the Cmax for the methylphenidate and CBD arm to the methylphenidate and placebo arm of each subject.
Arm/Group | All Participants
Number analyzed (Participants) | 24
Ratio | 1.08 [0.85 to 1.37]

2. Primary Outcome: Differences in the Geometric Mean Ratio (GMR) of the Area Under the Time Curve 0-infinity (AUCinf) for Methylphenidate Will be Compared Between the Two Exposure Conditions; i.e. Methylphenidate + CBD vs Methylphenidate + Placebo.
Description: All methylphenidate plasma concentrations were quantified using liquid-liquid extraction method and LC-MS/MS analysis. The terminal elimination rate constant (λz) was estimated by linear least-squares regression of the terminal portion of the plasma concentration (on natural logarithmic scale)-time curve. The area under the plasma concentration-time curve of methylphenidate AUC 0-8h were calculated according to the linear trapezoidal rule. AUC8-inf was extrapolated by using the last observed concentration of MPH (Clast) and dividing it by λz. AUC0-8 was added to AUC8-inf to get AUCinf. The GMR of the AUCinf for MPH were compared between the two exposure conditions, i.e., MPH with CBD versus MPH with placebo. In brief, if the 90% confidence interval (CI) of GMR for Cmax between the CBD group and placebo group was beyond the FDA's established bioequivalent limits of 0.8-1.25, the result was interpreted to represent a DDI. A GMR greater than 1.25 would be indicative of a DDI.
Time Frame: 0-8 hours (determined), 8 hours-infinity (extrapolated)
Population: Each subject served as their own control, so since all 12 subjects that completed the study went through both arms, we were able to analyze the both arms for each subject. Hence, 12 subjects gave us 24 arms (2 arms/subject). The AUCinf for each subject in the methylphenidate and CBD arm was directly compared to their methylphenidate and placebo arm, allowing us to determine the ratio of change in the presence of CBD.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Groups:
- All Participants: Methylphenidate and CBD Arm Only
  Subjects received a three day run in of CBD 750 mg orally twice daily (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]). On day four, all subjects returned to the clinical research center to receive one oral dose of CBD 750 mg orally (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
  Methylphenidate and Placebo Arm Only
  Subjects received a three day run in of 7.5 ml of Epidiolex® placebo solution (no CBD) orally twice daily. On day four, all subjects returned to the clinical research center to receive one oral dose of 7.5 mL of Epidiolex® placebo solution (no CBD) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
  The subsequent analysis compared the geometric mean ratio of the AUC for the methylphenidate and CBD arm to the methylphenidate and placebo arm of each subject.
Arm/Group | All Participants
Number analyzed (Participants) | 24
Ratio | 1.09 [0.89 to 1.32]

3. Other Pre Specified Outcome: Peak Methylphenidate Plasma Concentration (Cmax) for Methylphenidate and CBD Arms and Methylphenidate and Placebo Arms.
Description: Plasma methylphenidate (MPH) concentrations for both arms were determined by using a liquid-liquid extraction method and LC-MS/MS analysis. Peak concentration (Cmax) was reported as observed for each subject (highest observed plasma concentration of methylphenidate).
Time Frame: 8 hours
Population: Each subject served as their own control, so since all 12 subjects that completed the study went through both arms, we were able to analyze the both arms for each subject. Hence, 12 subjects gave us 24 arms (2 arms/subject). The Cmax for each subject in the methylphenidate and CBD arm and the methylphenidate and placebo arm was directly reported/analyzed below.
Measure: Mean (Full Range); unit: ng/mL
Groups:
- Methylphenidate and CBD Arm Only: Subjects received a three day run in of CBD 750 mg orally twice daily (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]). On day four, all subjects returned to the clinical research center to receive one oral dose of CBD 750 mg orally (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
- Methylphenidate and Placebo Arm Only: Subjects received a three day run in of 7.5 ml of Epidiolex® placebo solution (no CBD) orally twice daily. On day four, all subjects returned to the clinical research center to receive one oral dose of 7.5 mL of Epidiolex® placebo solution (no CBD) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
Arm/Group | Methylphenidate and CBD Arm Only | Methylphenidate and Placebo Arm Only
Number analyzed (Participants) | 12 | 12
ng/mL | 13.5 [6.9 to 26.5] | 12.2 [6.6 to 22.8]

4. Other Pre Specified Outcome: Time to Peak Methylphenidate Plasma Concentration (Tmax) for Methylphenidate and CBD Arms and Methylphenidate and Placebo Arms.
Description: Plasma methylphenidate (MPH) concentrations for both arms were determined by using a liquid-liquid extraction method and LC-MS/MS analysis. The time to peak plasma methylphenidate concentrations (Tmax) was reported as observed for each subject.
Time Frame: 8 hours
Population: Each subject served as their own control, so since all 12 subjects that completed the study went through both arms, we were able to analyze the both arms for each subject. Hence, 12 subjects gave us 24 arms (2 arms/subject). The Tmax for each subject in the methylphenidate and CBD arm and the methylphenidate and placebo arm was directly reported/analyzed below.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Methylphenidate and CBD Arm Only | Methylphenidate and Placebo Arm Only
Number analyzed (Participants) | 12 | 12
hours (h) | 1.25 [0.5 to 3] | 1.75 [0.5 to 3]

5. Other Pre Specified Outcome: Area Under the Time Curve 0-8hours (AUC0-8h) for Methylphenidate for the Two Exposure Conditions; Methylphenidate and CBD and Methylphenidate and Placebo.
Description: All methylphenidate plasma concentrations were quantified using liquid-liquid extraction method and LC-MS/MS analysis. The area under the plasma concentration-time curve of methylphenidate AUC 0-8h was calculated according to the linear trapezoidal rule.
Time Frame: 8 hours
Population: Each subject served as their own control, so since all 12 subjects that completed the study went through both arms, we were able to analyze the both arms for each subject. Hence, 12 subjects gave us 24 arms (2 arms/subject).
Measure: Mean (Full Range); unit: ng/mL*h
Arm/Group | Methylphenidate and CBD Arm Only | Methylphenidate and Placebo Arm Only
Number analyzed (Participants) | 12 | 22
ng/mL*h | 55.7 [31.6 to 80.7] | 49.6 [30.7 to 74.3]

6. Other Pre Specified Outcome: Area Under the Time Curve 0-infinity (AUCinf) for Methylphenidate for the Two Exposure Conditions for Methylphenidate and CBD and Methylphenidate and Placebo.
Description: All methylphenidate plasma concentrations were quantified using liquid-liquid extraction method and LC-MS/MS analysis. The terminal elimination rate constant (λz) was estimated by linear least-squares regression of the terminal portion of the plasma concentration (on natural logarithmic scale)-time curve. The area under the plasma concentration-time curve of methylphenidate AUC 0-8h were calculated according to the linear trapezoidal rule. AUC8-inf was extrapolated by using the last observed concentration of MPH (Clast) and dividing it by λz. AUC0-8 was added to AUC8-inf to get AUCinf.
Time Frame: 0-8 hours (determined), 8 hours-infinity (extrapolated)
Population: as for outcome 5
Measure: Mean (Full Range); unit: ng/mL*h
Arm/Group | Methylphenidate and CBD Arm Only | Methylphenidate and Placebo Arm Only
Number analyzed (Participants) | 12 | 12
ng/mL*h | 70.7 [38.6 to 103.3] | 63.6 [42.6 to 98.6]

7. Other Pre Specified Outcome: Half Life Determination (t1/2) for Methylphenidate for the Two Exposure Conditions for Methylphenidate and CBD and Methylphenidate and Placebo.
Description: All methylphenidate plasma concentrations were quantified using liquid-liquid extraction method and LC-MS/MS analysis. The terminal elimination rate constant (λz) was estimated by linear least-squares regression of the terminal portion of the plasma concentration (on natural logarithmic scale)-time curve. The elimination half-live (t1/2) was then calculated using the formula t1/2 = 0.693/λz.
Time Frame: 8 hours
Population: as for outcome 5
Measure: Mean (Full Range); unit: hours (h)
Arm/Group | Methylphenidate and CBD Arm Only | Methylphenidate and Placebo Arm Only
Number analyzed (Participants) | 12 | 12
hours (h) | 3.17 [2.24 to 4.52] | 3.12 [1.76 to 4.54]

ADVERSE EVENTS:
Time Frame: Subjects participation lasted 45 days
Groups:
- Methylphenidate and CBD Arms Only: Subjects received a three day run in of CBD 750 mg orally twice daily (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]). On day four, all subjects returned to the clinical research center to receive one oral dose of CBD 750 mg orally (administered as as 7.5 mL of Epidiolex® solution [100 mg/ml]) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
- Methylphenidate and Placebo Arms Only: Subjects received a three day run in of 7.5 ml of Epidiolex® placebo solution (no CBD) orally twice daily. On day four, all subjects returned to the clinical research center to receive one oral dose of 7.5 mL of Epidiolex® placebo solution (no CBD) and one 10 mg tablet of dl-methylphenidate (Ritalin®) orally in a fed state (a 30 minute standardized breakfast).
Arm/Group | Methylphenidate and CBD Arms Only | Methylphenidate and Placebo Arms Only
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 1/14 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate and CBD Arms Only (N=14) | Methylphenidate and Placebo Arms Only (N=12)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT04603391/Prot_SAP_001.pdf